CLINICAL TRIAL: NCT06133439
Title: Implementing Evidence Based Colorectal Cancer Screening in Rural Clinics
Brief Title: Rural Indiana Screening for Colorectal Cancer
Acronym: RISCC
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Melvin and Bren Simon Cancer Center (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Victoria L. Champion, Professor, Indiana University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: 15956; R01CA276659 (NIH)
Record Dates: First submitted 2023-11-06; First posted 2023-11-15 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Intervention Model Description: Cluster-Randomized Stepped Wedge design. Clinics will be randomized to one of three clusters that include four defined phases each consisting of nine-month segments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Phase 1 (No Intervention): Usual care and planning period.
- Phase 2 (Other): Implementation period.
  Clinics are randomized into clusters
  Interventions: Behavioral: Colorectal Screen rates with implementation of evidence-based intervention
- Phase 3 (Other): Maintenance period.
  Interventions: Behavioral: Colorectal Screen rates with implementation of evidence-based intervention

INTERVENTIONS:
Behavioral: Colorectal Screen rates with implementation of evidence-based intervention — Mailed FIT kits, Cologuard, and diagnostic colonoscopies.
  Arms: Phase 2; Phase 3

SUMMARY:
The goal of this implementation study is to support an evidence-based intervention to the improve colorectal cancer (CRC) screening and diagnostic colonoscopy rates in rural Indiana. The main questions the study aims to answer are:

* How does the implementation of an evidence based intervention to increase CRC screening in rural Indiana improve CRC screening and diagnostic colonoscopy rates, defined as completed screening episode?
* Will dose and type of implementation strategies contribute to differences in contextual factors and readiness as well as different levels of implementation outcomes (reach and implementation) in rural clinic?
* Will Contextual factors (innovation, recipient, inner and outer context) and implementation outcomes (reach, and implementation) vary with the levels of CRC screening and diagnostic colonoscopy following active implementation (effectiveness) and throughout maintenance compared to baseline (usual care)?
* What is the cost and budget impact of the deployment of implementation strategies and processes for rural clinics and evaluate the cost-effectiveness of implementing and sustaining the CRC screening intervention?

Approach: Participating clinics tasks consist of mailing FIT kits, sending text messages, phone reminders, and the use of a Patient Navigator to initiate a screening episode with eligible patients who are 45-75 (and have no colonoscopy in the last 10 years or FIT in the last 12 months) as identified from medical records.

DETAILED DESCRIPTION:
In Aim 1, the investigators will evaluate the ability of an implementation of an EBI to improve CRC screening and diagnostic colonoscopy rates, defined as completed screening episode (effectiveness) through implementation of an EBI for CRC screening in rural Indiana. The investigators hypothesize that a complete screening episode of CRC screening (FIT or screening colonoscopy), including diagnostic colonoscopy uptake following positive FIT, will be higher following implementation of an EBI and throughout maintenance compared to baseline (usual care). Resolution with diagnostic colonoscopy and repeat screening with FIT will be handled as exploratory outcomes.

In Aim 2, the investigators will evaluate the variation in contextual factors (innovation, recipient, inner and outer context), implementation strategies and implementation outcomes (reach and implementation) using mixed data (qualitative interviews and quantitative measures) to build implementation profiles of nine rural clinics.

In Aim 3, the investigators estimate the cost and budget impact of the deployment of implementation strategies and processes for rural clinics and evaluate the cost-effectiveness of implementing and sustaining the CRC screening intervention.

Study Overview: The investigators will partner with the IRHA, a not-for-profit organization, that was founded in 1997 to meet the healthcare needs of rural residents including Medicare and Medicaid recipients in underserved areas in Indiana. Nine IRHA with CRC screening rates below the state average of 68% were selected.

Approach and Design: The EBI for CRC screening consists of mailing an opportunity for patients not up to date with CRC screening to obtain a colonoscopy, Cologuard or FIT kit. Patients are provided with an opportunity to talk to a patient navigator and select screening options. Risk status for colorectal cancer is assessed. To initiate a screening episode, screening eligible patients who are 45-75 (no colonoscopy in the last 10 years or FIT in the last 12 months) will be identified from medical records

A centralized PN will serve all clinics during implementation, but this role will transition to clinic staff during maintenance. The PN will provide support to patients making decisions about the correct CRC screening test, scheduling a screening colonoscopy, and follow-up with a diagnostic colonoscopy when an FIT is positive.43,57-71 A standard operating procedure (SOP) will be developed during planning to support the navigation protocol and the transition of the PN role to clinic staff during maintenance. Navigation may include further assessment or confirmation of risk status, discussion about CRC screening or scheduling of a screening colonoscopy. With verbal consent, all calls will be recorded. Using the SOP, clinic staff who have basic medical assistant training will be able to support navigation when the PN role is transitioned to the clinic. A fidelity checklist will be used to assess 25% of all recorded calls for consistency in delivering the navigation protocol.

A positive stool-based test will prompt a stepped approach to counseling for diagnostic colonoscopy.

Implementation Strategy: The implementation strategy includes four components: 1) external facilitation, 2) CC identification and preparation, 3) establishment of a collaborative learning environment and 4) promotion of local adaptation.

Implementation Process: Startup activities occur in Year 1 and include ordering materials and supplies, hiring and training staff, establishing monthly research team meetings and EAB meetings, refining data collection measures and meeting with consultants. Using input from clinic staff, the investigators will hire and train interviewers and establish processes for all data collection including computer interfaces and database management. A PN will be available in each clinic to counsel patients. During Phase 1, investigators will assess CRC screening rates and promotion/education activities to identify a baseline as well as determine costs associated with any currently implemented strategies. Phase 2 begins as each cluster is stepped into the implementation design. A CC will be selected at each clinic and a learning collective will be developed to inform and engage all clinic staff. Before developing a clinic-specific plan, the investigators will assess contextual factors by collecting data from clinic staff and patients to inform the implementation plan. Assessment of contextual factors will provide information about the evidence surrounding the EBI, motivation or self-efficacy of staff/patients for implementing the EBI and factors in the inner or outer context that would facilitate or present challenges to implementation.

Following assessment, the clinics will begin development of a plan to support the steps necessary to implement the EBI, including the need for resources such as technical support for EMR programming and development of computerized logs for use in tracking activities. The clinic-specific plan will be developed in partnership with the CC and clinic staff. The learning collaborative will inform the implementation plan development, educate staff about the implementation process, and identify areas where adaptations to the plan are needed. After planning, the clinics will execute the implementation plan. Computerized clinic logs will track all steps of implementing the intervention including FIT and Cologuard distribution and retrieval, scheduling, completion of colonoscopy (screening and diagnostic) and PN calls. During active implementation, both the EIS and CC will use tracking sheets to record all actions, and fidelity will be monitored monthly. Adaptations to the initial implementation plan will be carefully documented.

Phase 3 (Maintenance) follows active implementation and is used to monitor continued adoption of the EBI and subsequent CRC screening, including annual repeat FIT screening for those who completed an initial negative FIT and diagnostic colonoscopy following a positive FIT. Cost effectiveness of implementation will be measured.

ELIGIBILITY:
Inclusion Criteria:

* All participants will be staff employed at the respective clinics. Patients will be age 45 to 75 and either male or female. Age limitations are necessary because colorectal cancer screening doesn't start until 45 and ends at 75.

Exclusion Criteria:

* Under surveillance (inherited familial syndromes),history of inflammatory bowel disease, and a previous adenomatous polyp, or previous colorectal cancer.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 11 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Effectiveness and Maintenance | Up to 12 months
  The primary effectiveness measure will be the rate of uptake of a complete episode CRC screening, a rate that includes resolution of a positive FIT test with diagnostic colonoscopy.
Contextual factors | Up to 12 months
  Contextual factors will be measured at the beginning of Phase 2 and during the midpoint and end of Phase 3. Semi structured items are used for contextual factors and are guided by the iPARIHS framework. The final contextual factor construct assessed during the interview will be readiness to engage in implementation of the EBI, measured by the Organizational Readiness to Change Assessment (ORCA).
Implementation outcomes | Up to 36 months
  Measured by CC tracking forms, clinic logs that record all PN calls, adaptations to the implementation plan, fidelity measures and costs. The Clinic Implementation Tracking Form contains all essential tasks in the implementation plan including the dose and quality of intervention delivery. Overall quality of implementation and responsiveness to facilitation will be rated on a scale of 1 to 3. At the end of Phase 3, the investigators will interview two staff/clinic about their perceptions of the implementation. The investigators will also measure responses to a validated Acceptability scale using two staff/clinic at each clinic. All adaptations to the implementation plan will be recorded including rationale for change. Cost-data will be collected in phase 1 for usual care CRC screening promotion/education activities and throughout Phase 2 and 3 of implementation.

OTHER OUTCOMES:
Maintenance | Up to 36 month
  Maintenance will be assessed by interviewing clinic staff to determine if the EBI will be maintained, barriers and facilitators to EBI use, and adaptations made to the implementation process.

CONTACTS AND LOCATIONS:
Overall Officials: Victoria Champion, PhD, Principal Investigator — Indiana University
Locations (1):
- Monroe Family Medicine (Adams Medical Group Monroe), Monroe, Indiana, United States

IPD SHARING:
Plan to Share IPD: No